CLINICAL TRIAL: NCT04598763
Title: Evaluation of Two Methods of Olfactory Rehabilitation in Post-viral Loss of Smell: Classic and Intensive
Acronym: Odorat-Covid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020PI098
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-07

CONDITIONS: Olfaction Disorders
MeSH Terms: conditions — Olfaction Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classic group (Other): the "classic" group receives classic olfactory rehabilitation using 4 scents most used in the literature (rose, eucalyptus, lemon, clove)
  Interventions: Other: smell the odors of the olfactory rehabilitation kit according to the classic or intensive method
- intensive (Other): the "intensive" group receiving olfactory rehabilitation using 8 scents (rose, eucalyptus, lemon, cloves, strawberries, cut grass, lavender, spruce).
  Interventions: Other: smell the odors of the olfactory rehabilitation kit according to the classic or intensive method

INTERVENTIONS:
Other: smell the odors of the olfactory rehabilitation kit according to the classic or intensive method — regardless of the randomization group, the patient will smell each odor for 10 seconds with a 10 second interval between odors.

SUMMARY:
One of the most common causes of loss of smell is upper respiratory tract infection. These disorders can be quantitative (hyposmia or anosmia) or qualitative (parosmia or phantosmia). Loss of smell has been found as a major and frequent clinical sign of Sars Cov2 infection (more than 50% of patients screened at the CHU Nancy). Spontaneous recovery remains possible. It usually occurs in the first month . But when symptoms persist, the therapeutic management of post-viral anosmias is poorly codified in the literature. Olfactory rehabilitation could allow faster recovery and better quality, but the published protocols are numerous and could only be tested on small inhomogeneous series of patients (mixture of post-viral and post-traumatic hypo-ansomy). The significant increase in the population of patients suffering from post-viral anosmia following the current pandemic situation makes it possible to consider a prospective study aiming to compare two olfactory rehabilitation protocols: "classic" and "intensive" in a population of patients. suffering only from post-viral hypoanosmia.

Hypothesis: Intensive or classic olfactory rehabilitation allows better results than spontaneous recovery

DETAILED DESCRIPTION:
80 patients will be recruited from among the patients consulting the otorhinolaryngology department of the Nancy CHRU for the assessment of viral post-infectious olfactory disorders.

The inclusion visit will be carried out during a standard routine care consultation with the following:

* an endoscopic endonasal examination
* the olfactory assessment (evaluation of smell by self-assessment, Dynachron-olfaction questionnaire, olfactory test by Sniffin 'Stick)

At the end of this assessment and after having received the information on the study and signed the consent form, the patients confirmed to be hypo-anosmic will then be randomized into 2 groups:

* "classic" olfactory rehabilitation group
* "intensive" olfactory rehabilitation group The rehabilitation kits (8 jars or 4 jars depending on the randomization group) will be provided to the patient with therapeutic education in their use.

The patient will carry out olfactory rehabilitation (intensive or classic) at home twice a day (morning and evening) for 32 weeks (i.e. 448 sessions). The patient will smell each odor for 10 seconds with an interval of 10 seconds between odors. Each training will be recorded by the patient in his olfactory rehabilitation agenda.

The patient will go again for a follow-up consultation for the renewal of his olfactory assessment at 4 months (follow-up visit 1) and at 8 months (follow-up visit 2) post-inclusion as part of the routine care of disorders of the smell post virus infection. In addition to the olfactory assessment during these visits, the investigator will also verify that the rehabilitation schedule is being kept.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient with a sudden loss of smell> 5 weeks linked to a viral infection (including SARS-CoV-2) of the upper respiratory tract treated in the ENT department of the CHRU Nancy
* Patient accepting olfactory rehabilitation
* Patient presenting with hyposmia or anosmia (confirmed by the threshold and identification tests of the Sniffin 'Stick kit)
* Patient affiliated to a social security scheme or beneficiary of such a scheme
* Patient who has received full research information and signed an informed consent.

Exclusion Criteria:

* Persons referred to in Articles L. 1121-5 to L. 1121-8 and L1122-2 of the Public Health Code:

Pregnant woman, parturient or nursing mother Person deprived of liberty by a judicial or administrative decision, Person undergoing psychiatric treatment under Articles L.3212-1 and L.3213-1 of the Public Health Code Minor (non-emancipated) Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice) Adult person unable to express consent and who is not the subject of a legal protection measure

* Qualitative smell disorder (cacosmia, hyperosmia, phantosmia, parosmia)
* Neurological, post-traumatic, neurodegenerative, congenital odor disorders
* Post-infectious loss of smell> 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
improvement in smell | eight month
  The change in smell is based on the comparison of the results of the olfactory assessment after / before olfactory rehabilitation obtained from a single method out of the three carried out:
  Sniffin 'Stick Test Results: Threshold Test Score and Actual Identification Test Score.
  TI score: sum of the individual scores of the threshold and identification measures (TI score varying from 0 to 32). It is used to classify patients in terms of normosmia, hyposmia and functional anosmia based on normative values of "Sniffin 'Sticks" (according to the age and sex of each subject) with the threshold at the tenth percentile of the database provided in the study published by Hummel and Kobal.
  Self-assessment by patients using a digital scale of smell, from 0 (no smell) to 10 (normal smell)
  Self-assessment using the Dynachron-olfaction questionnaire:each question is used to assess the patient's feelings about his discomfort in the nose using a scale from 0 (no discomfort) to 10 (unbearable

CONTACTS AND LOCATIONS:
Overall Officials: Duc Trung NGUYEN, Principal Investigator — CHRU de Nancy
Locations (1):
- CHRU de Nancy, Nancy, France